CLINICAL TRIAL: NCT06201949
Title: Efficacy of Articaine Infiltration in Anesthetizing Mandibular Second Primary Molars During Pulpotomy Procedure (Randomized Clinical Trial)
Brief Title: Articaine Infiltration in Anesthetizing Mandibular Second Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0636_2/2023
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Other: Articaine infiltration technique
- Control group (Active Comparator)
  Interventions: Other: Articaine nerve block technique

INTERVENTIONS:
Other: Articaine infiltration technique — infiltration will be performed with articaine and epinephrine 1/100 000 (Artinibsa, Inibsa, Barcelona, Spain) for all patients on their second pri-mary molar. The needle tip was placed in the buccal vestibule and then directed to the apex of the tooth and about one-third to one-fourth of the cartridge will be slowly discharged
  Arms: Test group
Other: Articaine nerve block technique — this technique will be performed with articaine and epinephrine 1/100 000 for all patients on their second primary molar with conventional technique inferior alveolar nerve block. The thumb will be placed on the occlusal surface of intended side and protruded toward the inner oblique ridge of ramus and then placed in touch with retromolar pad. The syringe will be directed between the two mandibular primary molars of opposite side and the needle will be pushed forward until hitting the bone, then the injection will be slowly done. After three to five minutes, treatment will be started, after numbness in the lower lip is achieved
  Arms: Control group

SUMMARY:
Background: Articaine hydrochloride has steadily grown in popularity, and studies have shown that articaine hydrochloride performs better than lidocaine due to an enhanced anes-thetic efficacy. The most common technique to anesthetize mandibular primary teeth is in-ferior alveolar nerve block (IANB) which induces a relatively sustained anesthesia and in turn may potentially traumatize soft-tissues. Therefore, the need of having an alternative technique of anesthesia with a shorter term but the same efficacy is reasonable.

Aim: Evaluating The effectiveness of Articaine infiltration versus conventional inferior al-veolar nerve block in anesthetizing the second primary mandibular molars during pulpoto-my procedure.

Materials and Methods: The study will be two-arm randomized controlled clinical trial, parallel design and it will be setup and reported according the CONSORT guidelines. A total of 52 healthy children aged 5-6 years, will be selected from Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Alexandria University, Egypt. Children will be selected with scores 3 or 4 according to Frankl behavioral rating scale. Each child selected will have at least one mandibular second primary molar that is indicat-ed for pulpotomy. Written informed consent will be obtained from guardian. Participants will be randomly and equally allocated to one of the two arms into two groups according to the technique of anesthesia that will be used.

Group I (Experimental group n =26) assigned to articaine infiltration anesthesia, while group II (Control group n = 26) assigned to the conventional IANB injection articaine.

Pain will be assessed by three diferent methods: physiological method using the Heart rate as vital parameter of pain, and will be recorded at base line, during injection, pulpotomy and stainless steel crown (SSC) preparation. Objective method using Sensory, Eye, Motor (SEM) scale, and subjective method where the pain will be evaluated by asking the child to express his experience using a modified face scale from the Maunuksela scale

ELIGIBILITY:
Inclusion Criteria:

* Positive or definitely positive behavior during preoperative assessments according to the Frankl's behavior ratings III and IV.
* Patients whose mandibular second primary molars are indicated for pulpotomy according to the AAPD.
* Patients whose parents will give their consent to participate

Exclusion Criteria:

* Children with any systemic disease or special health care.
* History of allergy to local anesthesia.
* Radiographic evidence of periapical or inter-radicular radiolucency
* Patients with previous negative dental experience.
* Presence of soft tissue lesions at the site of injection.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
change in heart rate | During procedure
  Heart rate (HR) is a physiological sign of pain.(30) It will be measured using a pulse oximeter.
change in pain level | During procedure
  Sound, Eye, Motor (SEM) Scale(31) (Appendix III), will used as an ob-jective method for pain assessment during LA administration, pulpo-tomy and SSC. It comprises the following parameters: (1) Sound, (2) Eye, (3) Motor. For each child, the sounds, eye symptoms and body movements will be evaluated independently by a blind impartial ob-server using the recorded video tapes. The slightest manifestation of the sound, eyes, or motion of the patient is graded in four levels: com-fort, mild, moderate, and severe discomfort, and subsequently given grades 1, 2, 3, 4, respectively. SEM score will be calculated by sum-ming the three grades of the parameters.

SECONDARY OUTCOMES:
Adevrse events | After 24 hours
  The presence of any adverse events including infection, oral/tooth pain, patients will be seen after 24 hours to detect any lip/cheek biting and parasethia

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt